CLINICAL TRIAL: NCT00122590
Title: Prospective Trial to Evaluate How Therapeutic Drug Monitoring of Protease Inhibitors Increases Virologic Success and Tolerance of HAART (ANRS 111 COPHAR2)
Brief Title: Evaluation of Therapeutic Drug Monitoring of Protease Inhibitors on Virologic Success and Tolerance of Highly Active Antiretroviral Therapy (HAART)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS111 COPHAR 2
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2005-08-01 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: protease inhibitors; nelfinavir; lopinavir; indinavir; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Indinavir; Ritonavir

INTERVENTIONS:
Drug: nelfinavir
Drug: lopinavir/r
Drug: indinavir
Drug: ritonavir

SUMMARY:
This Cophar2 study is a trial which evaluates repeated early therapeutic drug monitoring, from weeks 2 to 24, after the initiation of HAART including either indinavir/r, lopinavir/r or the new 625 mg formulation of nelfinavir twice-a-day (bid). If trough concentrations were out of the range given for each protease inhibitor (PI), the PI dose was adjusted.

DETAILED DESCRIPTION:
Because of the large pharmacokinetic inter-patient variability of protease inhibitors (PI), therapeutic drug monitoring (TDM) of protease inhibitor (PI) has been proposed to improve efficacy and tolerance of PI-containing HAART. The objective of the Cophar2 trial is to evaluate the feasibility and the impact of an early therapeutic drug monitoring in PI-naive HIV-1 infected patients in order to warrant virological success and safety of HAART.

It is a prospective, open, multicenter trial with repeated early TDM (weeks 2, 8 or 16, 24) after the initiation of HAART including either indinavir/r (IDV), lopinavir/r (LPV) or the new 625 mg formulation of nelfinavir (NFV) bid. It was planned to include 99 PI-naïve HIV-1 infected patients over 18 years old, 33 for each PI. Concentrations were measured by HPLC in each center. If trough concentrations were out of the range of 150-500, 2500-7000 or 1500-5500 ng/ml for IDV, LPV and NFV respectively, the PI doses were adjusted possibly more than once during the first 24 weeks of follow-up. Adjustments were done by steps of one pill (200, 133/33 or 250 mg for IDV, LPV/r or NFV, respectively) bid. Failure of the strategy was defined by either two consecutive viral loads over 200 copies/ml between weeks 16 and 48, or a validated PI-related adverse event grade III or IV or a grade II diarrhoea or renal lithiasis. Patients without adverse events before week 16 were defined as assessable if they had at least the virological assessment of week 16.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV-1
* Needing an antiretroviral treatment according to standard of care
* HIV viral load greater than 1000 copies/ml
* Beginning a treatment containing a PI (indinavir with or without ritonavir, nelfinavir, lopinavir + ritonavir) and 2 reverse transcriptase inhibitors
* PI-naive
* Antiretroviral treatment-naive or already treated with reverse transcriptase inhibitors but if the viral genotypic test does not show more than 2 major mutations (including T215Y/F, Q151M, M184V/I, V75M/S, L74V) and if 3 nucleoside analogues are still active except for didanosine.

Exclusion Criteria:

* Pregnant women and nursing mothers
* Acute HIV infection
* Diabetes
* Renal insufficiency with creatinine clearance below 30 ml/min
* Cardiac insufficiency
* Hepatic insufficiency with TP below 60%
* Treatment with known interactions with PI
* Chemotherapy against Kaposi's sarcoma, lymphoma, neoplasia
* Treatment containing interferon (INF) or interleukin-2 (IL2) or HIV- immune vaccine
* Treatment with hypolipemic drugs
* Laxative treatment
* Previous renal colic
* Diarrhoea with more than 5 stools/day since one week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115
Dates: Start 2002-07; Study Completion 2005-03

PRIMARY OUTCOMES:
treatment failure defined as viral load greater than 200 copies/ml between week 16 (W16) and week 48 (W48) (confirmed by 2 samples spiked at least 15 days apart but no more than 45 days after virological failure, assayed by 50 copies/ml method)
toxicity related to PI, defined as adverse event grade 3 or 4 with ANRS quotation, renal colic, diarrhoea grade 2, or cholesterolemia over 10 times the normal value

SECONDARY OUTCOMES:
virological failure: viral load over 200 copies/ml between W16 and W48 (confirmed by 2 samples spiked at least 15 days apart but no more than 45 days after virological failure, assayed by 50 copies/ml method)
toxicity related to PI: adverse events grade 3 or 4 with ANRS quotation, renal colic, diarrhoea grade 2, or cholesterolemia over 10 times the normal value
patients with trough plasma concentrations outside the therapeutic range at W24 and W48
concentration changes with dosage variation
time to obtain a viral load below 200 copies/ml
relationship between adverse events grade 3 or 4 related to PI and plasma concentration at week 2 (W2)
relationship between pharmacokinetic parameters and/or plasma concentrations and the drop of viral load between day 0 (D0) and W2 and between D0 and week 4 (W4)
relationship between pharmacokinetic parameters and viral mutations occurring during the treatment of patients with virological failure (over 1000 copies/ml after week 24 [W24])
PI pharmacokinetic parameter estimation and evaluation of variability
pharmacokinetic variability of nucleoside analogues at W2
intracellular concentration of nucleoside triphosphate derivatives at W2 (trough and maximum) and relationship between virological response and adverse events
relationship between inhibitory quotient of indinavir and virological response

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Salmon, MD, Principal Investigator — Service de Medecine Interne Hopital Cochin Paris; France Mentre, MD, Study Chair — Inserm EMI 03 57
Locations (1):
- Service de Medecine Interne Hopital Cochin, Paris, France